CLINICAL TRIAL: NCT06914934
Title: A 6-Month, Double-Blind, Placebo-Controlled Pilot Study of High-Dose Resveratrol in Patients With Stable Ischemic Heart Disease
Brief Title: Study of High-Dose Resveratrol in Patients With Stable Ischemic Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SW028
Record Dates: First submitted 2025-04-04; First posted 2025-04-07 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Ischaemic Heart Desease
Keywords: Supplements; Resveratol; Inflammation
MeSH Terms: conditions — Inflammation | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol arm (Experimental)
  Interventions: Dietary Supplement: High-dose resveratrol 500 mg/day
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: High-dose resveratrol 500 mg/day — High-dose resveratrol 500 mg/day (preferably a high-bioavailability formulation, e.g., trans-resveratrol with piperine or liposomal).
  Arms: Resveratrol arm
Other: Placebo — Placebo capsules, identical in appearance and schedule.
  Arms: Placebo

SUMMARY:
This 6-month, randomized, double-blind, placebo-controlled pilot study investigates whether high-dose resveratrol (500 mg/day), when added to standard therapy, can improve endothelial function and reduce inflammation in patients with stable ischemic heart disease. While preclinical data and small trials have shown promising effects on vascular health and inflammation, larger studies have lacked consistent results. This study aims to provide more robust clinical evidence by assessing flow-mediated dilation (FMD) and high-sensitivity C-reactive protein (hs-CRP) as primary outcomes in a well-defined patient group.

DETAILED DESCRIPTION:
This study is a 6-month, double-blind, placebo-controlled pilot randomized clinical trial designed to evaluate the effects of high-dose resveratrol (500 mg/day) on endothelial function and systemic inflammation in patients with stable ischemic heart disease (IHD). Despite widespread interest in resveratrol's cardioprotective potential, there remains limited high-quality clinical evidence supporting its benefit in established cardiovascular disease. Preclinical and small human studies suggest that resveratrol may enhance endothelial function via eNOS activation and oxidative stress reduction, reduce inflammation by lowering pro-inflammatory markers like CRP and cytokines, and mimic caloric restriction pathways through sirtuin activation. However, its clinical efficacy may be hindered by factors such as poor bioavailability, heterogeneous patient populations, and overlapping effects of standard cardiovascular drugs. This trial will randomize eligible participants, aged 45 to 75 with stable IHD and elevated inflammation or impaired endothelial function, to receive either resveratrol or placebo alongside their regular medication. The primary endpoints are changes in flow-mediated dilation (FMD) and high-sensitivity C-reactive protein (hs-CRP) from baseline to six months. Secondary outcomes include changes in inflammatory biomarkers, lipid profile, arterial stiffness, blood pressure, quality of life, and exercise tolerance. The study also assesses the safety and tolerability of long-term high-dose supplementation. With an estimated 70 participants (35 per arm), the study aims to detect a clinically meaningful 3% improvement in FMD with 80% power, contributing valuable data to guide future larger-scale investigations.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 45-75 years.
* Clinically documented stable ischemic heart disease (≥6 months post-myocardial infarction or post-revascularization).
* On stable, guideline-recommended cardiac medications (e.g., statins, beta-blockers, ACE inhibitors).
* Elevated hs-CRP (>2 mg/L) or impaired endothelial function (FMD <7%) at baseline (optional enrichment criterion).
* Able and willing to give written informed consent.

Exclusion Criteria:

* Heart failure with reduced ejection fraction <30% or New York Heart Association (NYHA) class III-IV.
* Severe hepatic or renal dysfunction.
* Decompensated diabetes (e.g., HbA1c >10%).
* Current or recent (past 3 months) use of high-dose antioxidant/anti-inflammatory supplements (other than a standard multivitamin).
* Known allergy or intolerance to resveratrol.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | 6 months
  Change in endothelial function: measured by brachial artery flow-mediated dilation from baseline to 6 months
Change in systemic inflammation | 6 months
  Change in systemic inflammation: measured by hs-CRP from baseline to 6 months

SECONDARY OUTCOMES:
Inflammatory cytokines change IL-6 | 6 months
Inflammatory cytokines TNF-α | 6 months
Total cholesterol change | 6 months
LDL change | 6 months
Triglycerides change mg/dl | 6 months
Arterial stiffness change | 6 months
  measured by pulse wave velocity
Quality of life Seattle Angina Questionnaire change | 6 months
Exercise tolerance 6-minute walk test change | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No